CLINICAL TRIAL: NCT03818087
Title: Elevate! : Improving Outcomes for Older Patients With Breast Cancer:a Longitudinal Cohort and Patient Engagement Study
Brief Title: Elevate! : An Elderly Breast Cancer Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Rachel Freedman, MD, MPH, Primary Investigator, Dana-Farber Cancer Institute
Other Study IDs: 18-634
Record Dates: First submitted 2018-12-19; First posted 2019-01-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tissue will be collected from participant's prior surgeries and procedures. Some participants undergoing breast surgery during the five years of participation may have a sample of fresh tissue taken for research purposes in the operating room. Blood will be collected at registration and at serial timepoints over a period of five years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elevate: Participants over the age of 70 years old with early-stage breast cancer will be recruited.
  Interventions: Behavioral: Observational cohort

INTERVENTIONS:
Behavioral: Observational cohort — Patients will be followed by collecting clinical data, biospecimens, and quality of life assessments over a period of five years from registration.

SUMMARY:
This study is focused on understanding how the investigators can improve upon breast cancer and health outcomes for older participants with breast cancer.

DETAILED DESCRIPTION:
This study is focused on understanding how the investigators can improve upon breast cancer and health outcomes for older participants with breast cancer, a group of participants who often have low risk cancers, but who may do worse than younger participants with the same kind of cancers. Researchers want to better understand the experiences, barriers, and changes in physical function older participants with breast cancer have.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older at the time of diagnosis (as indicated by the date of breast biopsy)
* No more than 67 patients (1/3) will be aged 70-74, with the remaining patients on study ages 75 or older
* Any gender is eligible
* Invasive, non-metastatic breast cancer at diagnosis
* Those with prior diagnoses of pre-invasive (DCIS) or invasive breast cancer are eligible as long as their current diagnosis is felt by the treating provider to represent a NEW non-metastatic primary invasive breast cancer (e.g. someone with a nodal recurrence from prior disease are not eligible but those with a new contralateral breast cancer 3 years after a first breast cancer would be eligible)
* Any breast cancer subtype is allowed
* Breast cancer-diagnosing biopsy within 90 days of enrollment
* Receiving or will receive medical oncology care (+/- surgical and radiation oncology treatments) at the participating center: DFCI/satellites and affiliate sites
* Patients must be able to understand, speak, and read English or assign a designated caregiver/proxy for the duration of the study who understands, speaks, and reads English and who is willing to assist with filling out the survey components which do not have a validated, translated version. This is because the surveys are not readily available in multiple languages as a whole, although some components (such as the Geriatric Assessment and PROs are readily available in multiple languages).
* If a patient scores 11 or higher on the baseline Orientation-Memory-Concentration Test done at baseline (Appendix E), a proxy/designee must then be assigned to help the patient fill out the questionnaires for the duration of the study in order to participate. The treating provider will also be notified about the cognitive impairment.
* Ability to provide informed consent

Exclusion Criteria:

* Pathological or clinical stage 0, IV disease
* Those with nodal or metastatic recurrences at the time of enrollment
* Unable to speak and read English AND no designee who speaks and reads English, as above
* Unable to provide informed consent

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Age 70 or older at the time of diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Adjuvant treatment recommendations | 7 years
  Report treatment recommendations made to patients enrolled on the cohort
Adherence to hormonal therapy | 7 years
  We will survey patients on adherence
Barriers to treatment and adherence | 7 years
  We will survey patients on the reasons for adherence and poor adherence
Treatment patterns by age and other characteristics | 7 years
  We will examine treatment receipt and patterns by subtype of disease

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Freedman, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Northern Light Cancer Care, Bangor, Maine
  - Brigham and Women Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lifespan Cancer Institute, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].